CLINICAL TRIAL: NCT07071688
Title: Predictive Value of Peripheral Blood CHI3L1 for Tumor Radiosensitivity: A Prospective and Retrospective Cohort Study
Brief Title: Study of Peripheral Blood CHI3L1 to Predict Tumor Response to Radiotherapy
Status: Not yet recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-292
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Tumor; Radiotherapy; Biomarker
Keywords: Tumor; Radiotherapy; Radioresistance; CHI3L1
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Radiotherapy is an important treatment for many malignant tumors. However, radioresistance remains a major cause of treatment failure, often leading to tumor recurrence or progression. As a key factor affecting prognosis, radioresistance currently lacks reliable methods for identifying high-risk individuals before treatment. Liquid biopsy, as a non-invasive and dynamic monitoring tool, offers unique advantages for real-time assessment. Previous studies from our group have shown that peripheral blood levels of CHI3L1 are significantly elevated in patients with radioresistant tumors and may serve as a predictive biomarker for radiotherapy sensitivity. This study aims to conduct a multicenter, bidirectional cohort study to systematically evaluate the predictive value of peripheral blood CHI3L1 as a pan-cancer biomarker for tumor response to radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent form;
* Age ≥ 18 years;
* No restrictions on sex;
* Histologically confirmed diagnosis of one of the following malignant tumors: nasopharyngeal carcinoma, head and neck cancer, lung cancer, breast cancer, gastric cancer, colorectal cancer, glioma, esophageal cancer, liver cancer, cholangiocarcinoma, cervical cancer, prostate cancer, or bladder cancer;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.

Exclusion Criteria:

* Patients with any serious comorbidities that may pose an unacceptable risk or adversely affect compliance with the study protocol. Examples include unstable heart disease requiring treatment, chronic hepatitis, renal disease with poor clinical status, uncontrolled diabetes mellitus (fasting blood glucose > 1.5 × ULN), or psychiatric disorders.
* Deemed unsuitable for participation in the study at the discretion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with tumors who require radiotherapy
Sampling Method: Probability Sample
Enrollment: 338 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | Through study completion, up to 3 years
  Objective Response Rate (ORR) after Radiotherapy in Tumor Patients

SECONDARY OUTCOMES:
Local Control Rate | Through study completion, up to 3 years
  Local Control Rate after Radiotherapy in Tumor Patients
Local Relapse Free Survival | Through study completion, up to 3 years
  Locoregional Recurrence-Free Survival after Radiotherapy in Tumor Patients
Progression Free Survival | Through study completion, up to 3 years
  Progression-Free Survival after Radiotherapy in Tumor Patients
Overall Survival | Through study completion, up to 3 years
  Overall Survival after Radiotherapy in Tumor Patients

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Nanfang hospital, Southern medical university, Guangzhou, Guangdong 510515, Guangzhou, Guangzhou
  - Huizhou Central People's Hospital, Huizhou, Huizhou
  - Meizhou People's Hospital, Meizhou Academy of Medical Sciences Meizhou, Meizhou,, Meizhou

IPD SHARING:
Plan to Share IPD: No